CLINICAL TRIAL: NCT01630668
Title: Efficacy of a One-a-Day L. Reuteri NCIMB 30242 Probiotic Supplement Capsule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Micropharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-12LCHM
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-a-Day L. reuteri NCIMB 30242 supplement capsule (Experimental)
  Interventions: Dietary Supplement: One-a-Day L. reuteri NCIMB 30242 supplement capsule
- One-a-Day placebo capsule (Placebo Comparator)
  Interventions: Dietary Supplement: One-a-Day placebo capsule

INTERVENTIONS:
Dietary Supplement: One-a-Day L. reuteri NCIMB 30242 supplement capsule — Once per day, 12 weeks
  Arms: One-a-Day L. reuteri NCIMB 30242 supplement capsule
Dietary Supplement: One-a-Day placebo capsule — Once per day, 12 weeks
  Arms: One-a-Day placebo capsule

SUMMARY:
Background: In recent years, probiotics have shown promise in treating a variety of diseases. Previously, the investigators have reported on the clinical efficacy of Lactobacillus reuteri NCIMB 30242 in improving the lipid profile in hypercholesterolemic adults.

Objective: The purpose of the study is to determine the lipid lowering efficacy of a One-a-Day probiotic supplement capsule containing Lactobacillus reuteri NCIMB 30242 over 12 weeks in subjects with hypercholesterolemia.

Design: The study design is a double-blinded, placebo-controlled, randomized, parallel-arm, multi-centre study. The study will last a total of 14 weeks, including a 2-week run-in period and a 12-week intervention period.

ELIGIBILITY:
Inclusion criteria:

* Males and females, aged 20 to 75 years (bounds included).
* LDL-C ≥ 3.40 mmol/L (<15% variation between visits V0 and V2-1).
* TG < 4.00 mmol/L (confirmed at visits V0 and V2-1).
* BMI range will be 23.0 to 32.5 kg/m2 (bounds included).
* Subject understands and accepts to follow the dietary recommendations advisable for hypercholesterolemic patients (according to NCEP-ATP III guidelines).
* Judged by the investigators as compliant (>80%) with product consumption (check at V2-1), and motivated.
* Signed informed consent form prior to inclusion in the study.
* Note: Subjects will be permitted to take stable doses of thyroid hormone and anti-hypertensive agents, as long as these are continued equivalently throughout the duration of study.
* If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation). OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:

  * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
  * Intrauterine devices
  * Vasectomy of partner
  * Total abstinence

Exclusion criteria:

* Use of cholesterol lowering prescription drugs within the last 6 months.
* Use of plant sterols, omega 3, fish oil, soy protein, soluble oat fiber, psyllium seed husk, or other cholesterol lowering non-prescription supplements within last 1 month.
* History of chronic use of alcohol (> 2 drinks/d).
* History of heavy smoking (≥ 20 cigarettes/d).
* Use of systemic antibodies, corticosteroids, androgens, or phenytoin.
* Immune-compromised subjects (e.g. AIDS, lymphoma, subjects undergoing long-term corticosteroid treatment)
* Subject having experienced any cardiovascular event (Myocardial infarction, coronary artery bypass, or other major surgical procedures) in the last 6 months.
* Subjects with elevated LDL-C (≥ 3.40 mmol/L) and high (>20%) CVD risk estimated by the Framingham risk score.
* Previously diagnosed Type I or Type II diabetes.
* Subject receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters.
* Subject currently involved in a clinical trial or in an exclusion period following participation in another clinical trial.
* History of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year).
* Clinically significant abnormal laboratory results at screening.
* Chronic user of probiotics or fibre laxative (greater than 2 doses/wk), or stimulant laxatives.
* History of eating disorders.
* Exercise greater than 15 miles/wk or 4,000 kcal/wk.
* For female subjects: Pregnancy, breast feeding, or intent to get pregnant.
* Allergy or sensitivity to test product ingredients
* Allergy or sensitivity to all 3 antibiotics (Clindamycin, Erythromycin and Ampicillin).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in serum LDL-cholesterol from baseline to endpoint between control and treatment groups. | Week 0 and Week 12 of intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada